CLINICAL TRIAL: NCT06715436
Title: The Effects of Ketogenic Diet Therapy Versus the Mediterranean Diet on Quality of Life in a Group of Patients With Multiple Sclerosis - the KETOMED-MS Study
Brief Title: Multiple Sclerosis and the Effects of Ketogenic Diet Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Collaborators: University of Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KETOMED-MS-2024
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; Ketogenic Dietary Therapy; Mediterranean diet
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Diet, Mediterranean; Diet, Ketogenic; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mediterranean Diet (Other): The MedDiet will be planned according to the Mediterranean diet pyramid. Energy prescriptions will be tailored to each patient's specific needs. The initial calorie prescription will be calculated taking into account usual dietary intake REE and physical activity level (PAL). Changes to calorie prescriptions will be made as needed during the course of follow-up. A minimum of 0.8-1 g of animal protein (e.g. eggs, milk, meat, poultry and fish) per kilogram of body weight per day will be given.
  Interventions: Dietary Supplement: Mediterranean Diet
- Ketogenic Diet (Experimental): Modified Atkins diet with a maximum of 20 g of carbohydrates per day. Fat-rich foods of plant origin will be encouraged in order to reach the prescribed daily caloric intake. Energy prescriptions will be tailored on each patient's specific requirements. The initial calorie prescription will be based on an average between the pre-diet intake, REE and physical activity levels. A minimum of 0.8-1 g of protein from animal sources (e.g. eggs, milk, meat, poultry and fish) per kilogram of body weight per day will be given.
  Interventions: Dietary Supplement: Ketogenic Diet
- Control group (Other): The control group will be asked to continue their dietary and lifestyle habits.
  Interventions: Dietary Supplement: Control group

INTERVENTIONS:
Dietary Supplement: Mediterranean Diet — The MedDiet will be planned according to the Mediterranean diet pyramid
  Arms: Mediterranean Diet
Dietary Supplement: Ketogenic Diet — Modified Atkins diet with a maximum of 20 g of carbohydrates per day.
  Arms: Ketogenic Diet
Dietary Supplement: Control group — The control group will be asked to continue their dietary and lifestyle habits
  Arms: Control group

SUMMARY:
Multiple sclerosis (MS) is an inflammatory and immune-mediated neurological disease with multifactorial etiology. The specific etiopathogenetic mechanisms of MS are still unknown but it is clear that it results from a combination of genetic and environmental factors. Several studies have reported the possible role of diet as a risk factor for MS and its progression. To date, many dietary patterns and their association with MS have been studied, but data is still limited and inconclusive. Mediterranean Diet (MedDiet) has been associated with a lower risk of developing MS, compared to a Western-style diet. In one of investigators' studies, higher MedDiet adherence was associated with a 6-fold greater likelihood of having lower disease severity than those with low adherence. A significant restriction of carbohydrates (up to ketogenesis) can have beneficial effects on various parameters (inflammatory markers, oxidative stress, altered glucose metabolism) which are altered in subjects with MS. Ketogenic diet therapies (KDTs) have been recommended mainly for children with drug-resistant epilepsy, but in recent years they have been applied to Multiple Sclerosis. Preclinical studies in animal models evaluating the efficacy of KDTs in experimental autoimmune encephalomyelitis (EAE) found a beneficial effect of diet in slowing of disease progression, improvement of motor disability, reduction of inflammatory cytokines and reactive oxygen species. In a randomized study, improvements in health-related quality of life (HRQL) scores and a slight decrease in EDSS scores were found. An open-label, single-arm study of 20 patients with RRMS also reported that, after 6 months of MAD, no subjects had new or enlarging FLAIR/T2 lesions, with a significant improvement in the EDSS score, the Modified Fatigue Impact Scale subscales and arm. A 3-arm parallel-arm randomized controlled pilot study was planned to determine the effectiveness of a modified Atkins diet (MAD) compared to a Mediterranean diet (MedDiet) on quality of life in a population with MS.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an inflammatory and immune-mediated neurological disease with multifactorial etiology. MS is one of the most important causes of disability in young adults and affects more women than men (with a male-female incidence ratio between 1.5:1 and 2.5:1). The specific etiopathogenetic mechanisms of MS are still unknown but it is clear that it derives from a combination of genetic and environmental factors. Several studies have reported the possible role of diet as a risk factor for MS and its progression. The possible role of dietary components on neuroinflammation, one of the main pathogenetic mechanisms of MS, has attracted a lot of interest. Diet and dietary components can be beneficial not only on MS symptoms but also on disease progression and disability status. To date, many dietary patterns and their association with MS have been studied, but the data is still limited and inconclusive. Notably, previous observational studies have found that MS patients tend to have a less healthy or more pro-inflammatory diet, compared to controls. Recently, Alfredsson and colleagues evaluated the risk of MS based on adherence to different dietary patterns (Western, Mediterranean and vegan/vegetarian diets). The authors reported that the Mediterranean Diet (MedDiet) was associated with a lower risk of developing MS, compared to a Western-style diet, while no significant associations were described between the vegetarian/vegan diet and the risk of MS. The positive association between MedDiet adherence and improved MS severity was recently confirmed by our study, in which high MedDiet adherence was associated with a 6-fold greater likelihood of having a lower severity of disease compared to those with low adherence to the MedDiet. Over the years, researchers have studied not only the neurological aspects of the disease but also the metabolic characteristics of MS patients. Insulin resistance, inflammatory markers, oxidative stress have been and are currently the main topics of interest. Studies have highlighted that MS is associated with altered glucose and insulin metabolism, which can negatively influence cognitive decline and dysfunction. All of these mechanisms can be modified through significant carbohydrate restriction that decreases glycemia and insulin levels and leads to ketogenesis. Dietary interventions aimed at inducing therapeutic ketosis are called ketogenic diet therapies (KDTs) and include different dietary regimes: the classic ketogenic diet (cKD), the medium chain triglyceride (MCT) diet, the modified Atkins diet (MAD). These protocols have been recommended mainly for children with drug-resistant epilepsy, but in recent years they have been applied to several other neurological pathologies such as Alzheimer's, Parkinson's and, recently, Multiple Sclerosis. Preclinical studies in animal models evaluating the efficacy of KDTs in experimental autoimmune encephalomyelitis (EAE) found a beneficial effect of diet. In particular, KDT slowed disease progression, improved motor disability, reduced inflammatory cytokines and reactive oxygen species. Choi et al. (2016) enrolled 60 patients with relapsing-remitting MS (RRMS) in a randomized, parallel 3-arm study to evaluate the safety and feasibility of a 6-month KDT or fasting-mimicking diets (FMD) on patients' quality of life. The study reported improvements in health-related quality of life (HRQL) scores of both the KDT group and the FMD group, at 3 and 6 months. Furthermore, a slight decrease in EDSS scores was reported in the FMD and KDT groups. An open-label, single-arm study tested a modified Atkins diet (MAD) for 6 months in a group of 20 patients with RRMS with the aim of evaluating the feasibility and safety of the diet. The study reported that, after 6 months of MAD, no subjects had new or enlarging FLAIR/T2 lesions, with significant improvement in EDSS score, Modified Fatigue Impact Scale (MFIS) subscales, and arm function (assessed through the Nine-Hole Peg Test). Similarly, in their phase II study, Brenton and colleagues confirmed their initial findings and described an improvement in depression (Beck Depression Inventory, BDI) and quality of life (Multiple Sclerosis Quality of Life-54, MSQoL -54).

Given this context, a 3-arm parallel-arm randomized controlled pilot study was planned to determine the effectiveness of a modified Atkins diet (MAD) compared to a Mediterranean diet (MedDiet) on quality of life, measured by the physical health subscale (CPH ) of MSQoL -54, in a population with MS followed at the Mondino Foundation Institute of Pavia, Italy. Safety, feasibility and general neurological, nutritional, motor and clinical outcomes were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing-remitting MS (RRMS) or progressive MS (PMS)
* Age between 18 and 60 years
* BMI between 18.5 kg/m2 and 39.9 kg/m2
* If on disease-modifying drugs, stable for 6 months, or no use of drugs in the previous 6 months
* Ability to give verbal and written consent

Exclusion Criteria:

* Patients actively engaged in a weight loss program or other specific diet (e.g. vegetarian, vegan); patients not willing to follow the assigned dietary pattern or patients with high adherence to MedDiet (MediLite score > 14)
* Pregnancy or breastfeeding
* Relapse or cortisone treatment within 30 days before study entry
* Clinically relevant metabolic, progressive or malignant diseases
* Intake of > 1 g/day of omega-3 fatty acid supplements
* Underweight (BMI<18.5 kg/m2) or severe obesity
* Significant cognitive-cooperative impairment
* Insulin-dependent diabetes mellitus (type I)
* Weight loss greater than 5 kg within 2 months prior to study entry
* Diagnosis or suspicion of an eating disorder
* Kidney stones
* Oral anticoagulant therapy
* Known alcohol and drug abuse

Telephonic interviews will be performed monthly to evaluate adherence to the dietary treatment and/or whether any changes in supplements use, physical activity, nutrition habits.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
The CPH subscale of the Multiple Sclerosis Quality of Life-54 (MSQoL -54) | Evaluation at baseline and after 6 months
  Quality of life will be assessed in terms of physical health referring to the CPH subscale of the MSQoL -54 after 6 months of treatment. ITS consists of 52 items grouped in 12 subscales plus two single items.
  All scores are transformed to scale from 0-100 and then added within each subscale to obtain the subtotal. By dividing the subtotal by the number of responses, the final score of the subscale is obtained. The scores final are in turn multiplied by a specific number at each subscale; adding the scores transformed in this way there is a value for "physical health" and one for "mental health". These two values, added, give the final score of the MSQoL-54. The higher scores demonstrate better HRQoL in patients.

SECONDARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | Evaluation at baseline and after 6 months
  Degree of disability, measured with the EDSS. Scores are based on examination by a neurologist, and climb by half unit increments from 0 to 10 as level of disability increases.They are based on the level of neurological impairment of eight functional systems in the brain: pyramidal, cerebellar, brainstem, sensory, bowel and bladder function, visual function, cerebral functions, other.
Multiple Sclerosis Functional Composite (MSFC) | Evaluation at baseline and after 6 months
  It is a 3-part, standardized, quantitative assessment instrument for use in clinical studies, particularly clinical trials, of multiple sclerosis: Timed 25-Foot Walk (T25W) for leg function and ambulation, 9-Hole Peg Test (9HPT) for arm and hand function, and Paced Auditory Serial Addition Test (PASAT-3) for cognitive function.
  For these instruments there are not the minimum and the maximum values. Execution time is calculated. Longer time corresponds to worse outcome.
Modified Fatigue Impact Scale (MFIS) | Evaluation at baseline and after 6 months
  This instrument provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The full-length MFIS consists of 21 items. MFIS total score can range from 0 to 84.
  MFIS score > 38 indicates moderate to severe fatigue.
The Pittsburgh Sleep Quality Index | Evaluation at baseline and after 6 months
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-report questionnaire that assesses sleep quality over a one-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score. Pittsburg scale's total score ranges from 0-21; where a higher score describes poorer sleep quality (score >5= inadequate sleep, score <5= adequate sleep)
The Beck Depression Inventory | Evaluation at baseline and after 6 months
  The inventory contains 21 self-report items which individuals complete using multiple choice response formats. It is composed of items relating to symptoms of depression such as hopelessness and irritability, cognitions such as guilt or feelings of being punished, as well as physical symptoms such as fatigue, weight loss, and lack of interest in sex. BDI score can vary from 0 to 63. A BDI score of < 9 is considered normal, a score of 11-16 mild mood disturbance, and 21-30 mild-moderate depression, >30 severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Tavazzi, MD, Principal Investigator — U.O. Sclerosi Multipla
Locations (1):
- U.O.Sclerosi Multipla, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alfredsson L, Olsson T, Hedstrom AK. Inverse association between Mediterranean diet and risk of multiple sclerosis. Mult Scler. 2023 Aug;29(9):1118-1125. doi: 10.1177/13524585231181841. Epub 2023 Jun 27. PMID 37366345
- [Background] Ascherio A. Environmental factors in multiple sclerosis. Expert Rev Neurother. 2013 Dec;13(12 Suppl):3-9. doi: 10.1586/14737175.2013.865866. PMID 24289836
- [Background] Ayromlou H, Hosseini S, Khalili M, Ayromlou S, Khamudchiyan S, Farajdokht F, Hassannezhad S, Amiri Moghadam S. Insulin resistance is associated with cognitive dysfunction in multiple sclerosis patients: A cross-sectional study. J Neuroendocrinol. 2023 Jun;35(6):e13288. doi: 10.1111/jne.13288. Epub 2023 Jun 15. PMID 37317829
- [Background] Azary S, Schreiner T, Graves J, Waldman A, Belman A, Guttman BW, Aaen G, Tillema JM, Mar S, Hart J, Ness J, Harris Y, Krupp L, Gorman M, Benson L, Rodriguez M, Chitnis T, Rose J, Barcellos LF, Lotze T, Carmichael SL, Roalstad S, Casper CT, Waubant E. Contribution of dietary intake to relapse rate in early paediatric multiple sclerosis. J Neurol Neurosurg Psychiatry. 2018 Jan;89(1):28-33. doi: 10.1136/jnnp-2017-315936. Epub 2017 Oct 9. PMID 28993476
- [Background] Black LJ, Rowley C, Sherriff J, Pereira G, Ponsonby AL, Lucas RM. A healthy dietary pattern associates with a lower risk of a first clinical diagnosis of central nervous system demyelination. Mult Scler. 2019 Oct;25(11):1514-1525. doi: 10.1177/1352458518793524. Epub 2018 Aug 7. PMID 30084751
- [Background] Brenton JN, Banwell B, Bergqvist AGC, Lehner-Gulotta D, Gampper L, Leytham E, Coleman R, Goldman MD. Pilot study of a ketogenic diet in relapsing-remitting MS. Neurol Neuroimmunol Neuroinflamm. 2019 Apr 12;6(4):e565. doi: 10.1212/NXI.0000000000000565. eCollection 2019 Jul. PMID 31089482
- [Background] Brenton JN, Lehner-Gulotta D, Woolbright E, Banwell B, Bergqvist AGC, Chen S, Coleman R, Conaway M, Goldman MD. Phase II study of ketogenic diets in relapsing multiple sclerosis: safety, tolerability and potential clinical benefits. J Neurol Neurosurg Psychiatry. 2022 Jun;93(6):637-644. doi: 10.1136/jnnp-2022-329074. Epub 2022 Apr 13. PMID 35418509
- [Background] Choi IY, Piccio L, Childress P, Bollman B, Ghosh A, Brandhorst S, Suarez J, Michalsen A, Cross AH, Morgan TE, Wei M, Paul F, Bock M, Longo VD. A Diet Mimicking Fasting Promotes Regeneration and Reduces Autoimmunity and Multiple Sclerosis Symptoms. Cell Rep. 2016 Jun 7;15(10):2136-2146. doi: 10.1016/j.celrep.2016.05.009. Epub 2016 May 26. PMID 27239035
- [Background] Esposito S, Bonavita S, Sparaco M, Gallo A, Tedeschi G. The role of diet in multiple sclerosis: A review. Nutr Neurosci. 2018 Jul;21(6):377-390. doi: 10.1080/1028415X.2017.1303016. Epub 2017 Mar 24. PMID 28338444
- [Background] International Multiple Sclerosis Genetics Consortium; Wellcome Trust Case Control Consortium 2; Sawcer S, Hellenthal G, Pirinen M, Spencer CC, Patsopoulos NA, Moutsianas L, Dilthey A, Su Z, Freeman C, Hunt SE, Edkins S, Gray E, Booth DR, Potter SC, Goris A, Band G, Oturai AB, Strange A, Saarela J, Bellenguez C, Fontaine B, Gillman M, Hemmer B, Gwilliam R, Zipp F, Jayakumar A, Martin R, Leslie S, Hawkins S, Giannoulatou E, D'alfonso S, Blackburn H, Martinelli Boneschi F, Liddle J, Harbo HF, Perez ML, Spurkland A, Waller MJ, Mycko MP, Ricketts M, Comabella M, Hammond N, Kockum I, McCann OT, Ban M, Whittaker P, Kemppinen A, Weston P, Hawkins C, Widaa S, Zajicek J, Dronov S, Robertson N, Bumpstead SJ, Barcellos LF, Ravindrarajah R, Abraham R, Alfredsson L, Ardlie K, Aubin C, Baker A, Baker K, Baranzini SE, Bergamaschi L, Bergamaschi R, Bernstein A, Berthele A, Boggild M, Bradfield JP, Brassat D, Broadley SA, Buck D, Butzkueven H, Capra R, Carroll WM, Cavalla P, Celius EG, Cepok S, Chiavacci R, Clerget-Darpoux F, Clysters K, Comi G, Cossburn M, Cournu-Rebeix I, Cox MB, Cozen W, Cree BA, Cross AH, Cusi D, Daly MJ, Davis E, de Bakker PI, Debouverie M, D'hooghe MB, Dixon K, Dobosi R, Dubois B, Ellinghaus D, Elovaara I, Esposito F, Fontenille C, Foote S, Franke A, Galimberti D, Ghezzi A, Glessner J, Gomez R, Gout O, Graham C, Grant SF, Guerini FR, Hakonarson H, Hall P, Hamsten A, Hartung HP, Heard RN, Heath S, Hobart J, Hoshi M, Infante-Duarte C, Ingram G, Ingram W, Islam T, Jagodic M, Kabesch M, Kermode AG, Kilpatrick TJ, Kim C, Klopp N, Koivisto K, Larsson M, Lathrop M, Lechner-Scott JS, Leone MA, Leppa V, Liljedahl U, Bomfim IL, Lincoln RR, Link J, Liu J, Lorentzen AR, Lupoli S, Macciardi F, Mack T, Marriott M, Martinelli V, Mason D, McCauley JL, Mentch F, Mero IL, Mihalova T, Montalban X, Mottershead J, Myhr KM, Naldi P, Ollier W, Page A, Palotie A, Pelletier J, Piccio L, Pickersgill T, Piehl F, Pobywajlo S, Quach HL, Ramsay PP, Reunanen M, Reynolds R, Rioux JD, Rodegher M, Roesner S, Rubio JP, Ruckert IM, Salvetti M, Salvi E, Santaniello A, Schaefer CA, Schreiber S, Schulze C, Scott RJ, Sellebjerg F, Selmaj KW, Sexton D, Shen L, Simms-Acuna B, Skidmore S, Sleiman PM, Smestad C, Sorensen PS, Sondergaard HB, Stankovich J, Strange RC, Sulonen AM, Sundqvist E, Syvanen AC, Taddeo F, Taylor B, Blackwell JM, Tienari P, Bramon E, Tourbah A, Brown MA, Tronczynska E, Casas JP, Tubridy N, Corvin A, Vickery J, Jankowski J, Villoslada P, Markus HS, Wang K, Mathew CG, Wason J, Palmer CN, Wichmann HE, Plomin R, Willoughby E, Rautanen A, Winkelmann J, Wittig M, Trembath RC, Yaouanq J, Viswanathan AC, Zhang H, Wood NW, Zuvich R, Deloukas P, Langford C, Duncanson A, Oksenberg JR, Pericak-Vance MA, Haines JL, Olsson T, Hillert J, Ivinson AJ, De Jager PL, Peltonen L, Stewart GJ, Hafler DA, Hauser SL, McVean G, Donnelly P, Compston A. Genetic risk and a primary role for cell-mediated immune mechanisms in multiple sclerosis. Nature. 2011 Aug 10;476(7359):214-9. doi: 10.1038/nature10251. PMID 21833088
- [Background] Jelinek GA, Hadgkiss EJ, Weiland TJ, Pereira NG, Marck CH, van der Meer DM. Association of fish consumption and Omega 3 supplementation with quality of life, disability and disease activity in an international cohort of people with multiple sclerosis. Int J Neurosci. 2013 Nov;123(11):792-800. doi: 10.3109/00207454.2013.803104. Epub 2013 Jun 3. PMID 23713615
- [Background] Katz Sand I. The Role of Diet in Multiple Sclerosis: Mechanistic Connections and Current Evidence. Curr Nutr Rep. 2018 Sep;7(3):150-160. doi: 10.1007/s13668-018-0236-z. PMID 30117071
- [Background] Keykhaei F, Norouzy S, Froughipour M, Nematy M, Saeidi M, Jarahi L, Amiri F, Malek Ahmadi M, Norouzy A. Adherence to healthy dietary pattern is associated with lower risk of multiple sclerosis. J Cent Nerv Syst Dis. 2022 May 6;14:11795735221092516. doi: 10.1177/11795735221092516. eCollection 2022. PMID 35558004
- [Background] Kobelt G, Thompson A, Berg J, Gannedahl M, Eriksson J; MSCOI Study Group; European Multiple Sclerosis Platform. New insights into the burden and costs of multiple sclerosis in Europe. Mult Scler. 2017 Jul;23(8):1123-1136. doi: 10.1177/1352458517694432. Epub 2017 Feb 1. PMID 28273775
- [Background] Kossoff EH, Zupec-Kania BA, Auvin S, Ballaban-Gil KR, Christina Bergqvist AG, Blackford R, Buchhalter JR, Caraballo RH, Cross JH, Dahlin MG, Donner EJ, Guzel O, Jehle RS, Klepper J, Kang HC, Lambrechts DA, Liu YMC, Nathan JK, Nordli DR Jr, Pfeifer HH, Rho JM, Scheffer IE, Sharma S, Stafstrom CE, Thiele EA, Turner Z, Vaccarezza MM, van der Louw EJTM, Veggiotti P, Wheless JW, Wirrell EC; Charlie Foundation; Matthew's Friends; Practice Committee of the Child Neurology Society. Optimal clinical management of children receiving dietary therapies for epilepsy: Updated recommendations of the International Ketogenic Diet Study Group. Epilepsia Open. 2018 May 21;3(2):175-192. doi: 10.1002/epi4.12225. eCollection 2018 Jun. PMID 29881797
- [Background] Martin-McGill KJ, Jackson CF, Bresnahan R, Levy RG, Cooper PN. Ketogenic diets for drug-resistant epilepsy. Cochrane Database Syst Rev. 2018 Nov 7;11(11):CD001903. doi: 10.1002/14651858.CD001903.pub4. PMID 30403286
- [Background] Uygun Ozel S, Bayram S, Kilinc M. The relationship between dietary profile and adherence to the Mediterranean diet with EDSS and quality of life in multiple sclerosis patients: a retrospective cross-sectional study. Nutr Neurosci. 2024 Apr;27(4):404-412. doi: 10.1080/1028415X.2023.2201026. Epub 2023 Apr 18. PMID 37071567
- [Background] Penesova A, Dean Z, Kollar B, Havranova A, Imrich R, Vlcek M, Radikova Z. Nutritional intervention as an essential part of multiple sclerosis treatment? Physiol Res. 2018 Aug 16;67(4):521-533. doi: 10.33549/physiolres.933694. Epub 2018 May 10. PMID 29750884
- [Background] Rouzitalab T, Shivappa N, Daneshzad E, Izadi A, Sanoobar M, Khandouzi N, Shiri-Shahsavar MR, Khalili M. Dietary patterns and risk of multiple sclerosis: Results of a double-center case-control study in Iran. Nutr Health. 2023 Sep;29(3):531-539. doi: 10.1177/02601060221082379. Epub 2022 Mar 2. PMID 35234101
- [Background] Stoiloudis P, Kesidou E, Bakirtzis C, Sintila SA, Konstantinidou N, Boziki M, Grigoriadis N. The Role of Diet and Interventions on Multiple Sclerosis: A Review. Nutrients. 2022 Mar 9;14(6):1150. doi: 10.3390/nu14061150. PMID 35334810
- [Background] Tredinnick AR, Probst YC. Evaluating the Effects of Dietary Interventions on Disease Progression and Symptoms of Adults with Multiple Sclerosis: An Umbrella Review. Adv Nutr. 2020 Nov 16;11(6):1603-1615. doi: 10.1093/advances/nmaa063. PMID 32504530
- [Background] Wahls TL. Dietary Approaches to Treating Multiple Sclerosis-Related Symptoms. Phys Med Rehabil Clin N Am. 2022 Aug;33(3):605-620. doi: 10.1016/j.pmr.2022.04.004. Epub 2022 Jun 25. PMID 35989054
- [Result] Guglielmetti M, Al-Qahtani WH, Ferraris C, Grosso G, Fiorini S, Tavazzi E, Greco G, La Malfa A, Bergamaschi R, Tagliabue A. Adherence to Mediterranean Diet Is Associated with Multiple Sclerosis Severity. Nutrients. 2023 Sep 16;15(18):4009. doi: 10.3390/nu15184009. PMID 37764792